CLINICAL TRIAL: NCT03382782
Title: Peer Navigators to Address Obesity-Related Concerns for African Americans With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois Institute of Technology (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); ACCESS Community Health Network (Other); Trilogy Inc. Behavioral Healthcare (Other)
Responsible Party: Principal Investigator, Patrick Corrigan, Distinguished Professor of Psychology, Illinois Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1U01MD010541 (NIH); 1U01MD010541 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Mental Disorder
Keywords: Obesity; Mental Disorder; Peer Navigator; Physical Health; Overweight; Serious Mental Illness
MeSH Terms: conditions — Obesity; Mental Disorders; Overweight | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Intervention Model Description: The behavioral weight loss intervention (BWLI) consists of an 8-month intervention phase followed by a 4-month maintenance phase. The initial intervention phase comprises four types of contact: 1) One-hour to one and a half hour group weight management class led by facilitator (once per week); 2) 45-minute physical activity class led by facilitator (1-2 per week); 3) 20-minute, individual visit with facilitator (once per month); 4) Weigh-in (once each week). Persons are randomly assigned to peer navigators to begin simultaneously with BWLI and run concurrently across the eight months of the intervention. PNs may work with participants to partner on BWLI homework, meet with participant and BWLI facilitator individually, attend health care appointments, and partner on tasks that arise out of those appointments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral Weight Loss Intervention (Active Comparator): Participants will enroll in the BWLI program for 12 months. BWLI consists of a 8-month initial intervention phase followed by 4-month maintenance phase. The initial intervention phase comprises four types of contact:
  * 1-hour to 1-hour, 30 minute group weight-management class led by facilitator (once per week; 26 classes followed by a one week break and an additional 8 weight management review classes)
  * 45 minute, physical activity led by facilitator (one-two times per week);
  * 20 minute, monthly individual visit with facilitator to address barriers to goals and appropriate skills; and
  * weigh-in during weight management group and individual visits (once each week).
  Interventions: Behavioral: BWLI
- BWLI & Peer Navigator (Experimental): Participants randomly assigned to this condition will begin simultaneously with BWLI and run concurrently across the eight months of the intervention. Peer navigators will meet individually and face-to-face with research participants in time and places convenient to the person as needed. Specific practices are determined by the research participant with the peer navigator and may include:
  * partnering with participant on BWLI homework;
  * meeting with participant and BWLI facilitator individually;
  * attending all other health care appointments; and
  * partnering on tasks that arise out of those appointments.
  Interventions: Behavioral: BWLI & Peer Navigator
- Integrated Care (Treatment as Usual) (Active Comparator): Participants in this arm will receive integrated care from their usual provider, which is treatment as usual. Integrated care is mental health specialty and general medical care providers working together to address the physical and behavioral health care needs of patients. One-third of research participants will be randomized to integrated care alone.
  Interventions: Behavioral: Integrated Care

INTERVENTIONS:
Behavioral: BWLI — BWLI includes group weight management classes, physical activity classes, individual sessions with a facilitator to address goals and barriers to weight loss, and weigh-ins.
  A punch card system will be implemented to incentivize participation for BHL classes. Each participant from the BWLI condition will be given a punch card, each punch card contains 10 spaces of punches, and will receive a punch at the end of each class (either BHL or physical activity) they attend. No punch will be given if they are more than 15 minutes late for BHL class or more than 5 minutes late for physical activity class. Participants can earn $5 per punch for up to $250. They will be allowed to cash in for $50 Visa gift card every 10 punches. They cannot cash in for a partially filled card. They must have the 10 full punches to cash in.
  Arms: Behavioral Weight Loss Intervention
Behavioral: BWLI & Peer Navigator — Participants receive the BWLI condition and partner with a peer navigator. Peer navigators will meet individually and face-to-face with participants to address their health and weight goals (i.e. working on BWLI homework, attending health care appointments, and facilitating diet and exercise activities). A punch card system will be implemented to incentivize participation for BHL classes. Each participant from BWLI & Peer Navigator will be given a punch card, each punch card contains 10 spaces of punches, and will receive a punch at the end of each class (either BHL or physical activity) they attend. No punch will be given if they are more than 15 minutes late for BHL class or more than 5 minutes late for physical activity class. Participants can earn $5 per punch for up to $250. They will be allowed to cash in for $50 Visa gift card every 10 punches. They cannot cash in for a partially filled card. They must have the 10 full punches to cash in.
  Arms: BWLI & Peer Navigator
Behavioral: Integrated Care — Participants receive integrated physical and mental health care from their usual provider.
  Arms: Integrated Care (Treatment as Usual)

SUMMARY:
People with serious mental illness such as schizophrenia and bipolar disorder experience high rates of physical illness and die earlier than people without serious mental illness (WHO, 2005). Health differences seem to be worse among African Americans (Weber, Cowan, Millikan & Niebuhr, 2009). High rates of obesity among this group contribute to health and wellness concerns (de Hert et al., 2011), with African American women at higher risk of obesity than men. Behavioral weight loss interventions (BWLIs) may promote diet and physical activity that lead to weight loss, but healthy food and safe physical activity options are less available in low-income neighborhoods. Peer navigators have been found to be effective in addressing health differences, and may help people living in low-income communities find healthy food and activity resources (Fischer, Sauaia, & Kutner, 2007). In addition, traumatic experiences are common among persons with serious mental illness as well as African Americans, and may impact weight.

Through this project, investigators will test two interventions designed to address overweight and obesity among African Americans with serious mental illness. The first is a BWLI designed for persons with serious mental illness and adapted to meet the needs of African Americans. This program has 8-month intervention phase and 4-month maintenance phase. The intervention includes group weight management classes, group physical activity, individual visits to address barriers to meeting weight goals, and weigh-ins. The second intervention is a peer navigator program that assists people with serious mental illness in meeting their health needs in the community. Two-hundred and seventy (270) research participants will be recruited and randomly assigned to one of three conditions: BWLI program, BWLI program plus peer navigator, and treatment as usual (integrated physical and mental health care). Investigators will evaluate these interventions over a 12-month period, and will track weight change, health behaviors, physical and mental health, recovery, and quality of life. Investigators also seek to understand the impact of gender and trauma on outcomes. Investigators hypothesize that peer navigators will improve outcomes over the BWLI program alone. Findings will advance knowledge and services to reduce racial disparities in obesity and comorbid health conditions for African Americans with serious mental illnesses.

DETAILED DESCRIPTION:
Persons with serious mental illness experience disproportionate rates of physical health morbidity and mortality (WHO, 2005). One reason is a metabolic syndrome marked by significant obesity which seems even worse for African Americans. Although research suggests behavioral weight loss interventions (BWLIs) may promote healthy lifestyle behaviors (diet and exercise) that leads to weight loss, these programs are hindered by several social determinants of health found in low-income communities with food and activity deserts that undermine program goals. Preliminary evidence finds that peer navigators (service providers in recovery from serious mental illness) can help people to better avail existing healthcare programs, thereby improving health. Based on this evidence, our community-based participatory research (CBPR) project develops and tests two existing interventions to address the weight concerns of African Americans with serious mental illness:

1. A BWLI developed for persons with serious mental illness (Goldberg et al., 2013) that will be evaluated for its responsiveness to the needs of African Americans with serious mental illness
2. A peer navigator program (PNP) (Corrigan et al., 2017) that assists people with serious mental illness in meeting their health needs in the community; the PNP will be adapted so peer navigators can augment the impact of BWLI in food and activity deserts.

As compared with men, African American women with serious mental illness are at an even higher risk for lifetime prevalence of obesity (Baskaran et al., 2014; Galletly et al., 2012). Through an administrative supplement, investigators have augmented the approach of our study to understand the role of gender on the attainment of weight goals, with a specific focus on trauma, an experience of particular importance to women's health.

Two-hundred and seventy (270) African Americans with serious mental illness who are overweight or obese will be randomized to one of three conditions after baseline assessments: integrated physical and mental health care, integrated physical and mental health care plus BWLI, or integrated physical and mental health care plus BWLI and peer navigator (PN).

The BWLI has a 8-month intervention phase followed by a 4-month maintenance phase. The intervention includes group weight management classes, physical activity, individual visits to address barriers to meeting goals and to develop skills, and weigh-ins. PNs will partner with participants on BWLI assignments, meet with participants and BWLI facilitators, or accompany participants to health care appointments and follow-up. In addition, PNs and participants will team up to assess community diet and activity resources, and based on this review, will develop strategies to address their diet and physical activity needs.

Investigators seek 70 participants per condition (N=210) to reach statistical power goals. Investigators will recruit 270 participants to account for expected loss-to-followup. Investigators will enroll participants in discrete cohorts every nine months.

Investigators will analyze fidelity, process, outcome and impact data, including the effect of BWLI and BWLI and PN on weight, waist circumference, blood pressure, health behavior, physical and mental health, recovery and quality of life. Measures will be repeated at 4, 8, and 12 months. To understand the impact of gender, investigators will stratify the sample on gender at recruitment and analyze all program outcome measures by gender. To better understand the impact of trauma, investigators will determine if trauma exposure moderates the effect of the study intervention. Investigators will also conduct post-hoc analyses to determine if gender matching between PNs and participants (e.g., female-female and male-male) led to better effects.

Investigators' main hypothesis is that the BWLI and PN condition will lead to greater weight loss and enhanced health behaviors compared with the two other conditions. Findings will advance knowledge and services to reduce racial disparities in obesity and comorbid health conditions for African Americans with serious mental illnesses.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Age 18 or older
* Serious mental illness (as indicated by disability)
* Identifies as either male or female
* Concerned about weight and health goals
* Willing to attend
* BMI of greater than or equal to 28

Exclusion Criteria:

* Currently receiving services from a peer support specialist or community health worker to work on weight-related goals
* Weigh more than 440 pounds
* Lifetime diagnosis of eating disorder
* Pregnant or plan to become pregnant
* Lifetime bariatric surgery
* No doctor permission for exercise
* Taking medication for weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must identify as female or male.
Enrollment: 234 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Corrigan, PsyD, Principal Investigator — Illinois Institute of Technology
Locations (3):
- United States (3):
  - Illinois Institute of Technology, Chicago, Illinois
  - Trilogy Behavioral Healthcare, Chicago, Illinois
  - Access Community Health Network, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Results will be available to researchers and service agencies, with quantitative data available from an expected 210 African American participants with serious mental illness who report concerns obesity or being overweight. No identifying information will be connected to the data and investigators do not believe that there is a possibility of deductive disclosure of subjects with unusual characteristics. Regardless, to ensure the protection of the human subjects involved in this research, investigators will make the data and associated documentation available to users only under a data-sharing agreement. Notice of available data will be posted in appropriate arenas including websites for the project: www.chicagohealthdisparities.org and www.ncse1.org.
Time Frame: Data will be available on 12-31-2020.
Access Criteria: To ensure the protection of the human subjects involved in our research, investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
URL: http://www.chicagohealthdisparities.org

REFERENCES:
- [Background] Baskaran A, Cha DS, Powell AM, Jalil D, McIntyre RS. Sex differences in rates of obesity in bipolar disorder: postulated mechanisms. Bipolar Disord. 2014 Feb;16(1):83-92. doi: 10.1111/bdi.12141. Epub 2013 Oct 29. PMID 24467470
- [Background] Corrigan PW, Kraus DJ, Pickett SA, Schmidt A, Stellon E, Hantke E, Lara JL. Using Peer Navigators to Address the Integrated Health Care Needs of Homeless African Americans With Serious Mental Illness. Psychiatr Serv. 2017 Mar 1;68(3):264-270. doi: 10.1176/appi.ps.201600134. Epub 2017 Jan 17. PMID 28093056
- [Background] DE Hert M, Correll CU, Bobes J, Cetkovich-Bakmas M, Cohen D, Asai I, Detraux J, Gautam S, Moller HJ, Ndetei DM, Newcomer JW, Uwakwe R, Leucht S. Physical illness in patients with severe mental disorders. I. Prevalence, impact of medications and disparities in health care. World Psychiatry. 2011 Feb;10(1):52-77. doi: 10.1002/j.2051-5545.2011.tb00014.x. PMID 21379357
- [Background] Fischer SM, Sauaia A, Kutner JS. Patient navigation: a culturally competent strategy to address disparities in palliative care. J Palliat Med. 2007 Oct;10(5):1023-8. doi: 10.1089/jpm.2007.0070. No abstract available. PMID 17985954
- [Background] Goldberg RW, Reeves G, Tapscott S, Medoff D, Dickerson F, Goldberg AP, Ryan AS, Fang LJ, Dixon LB. "MOVE!" Outcomes of a weight loss program modified for veterans with serious mental illness. Psychiatr Serv. 2013 Aug 1;64(8):737-44. doi: 10.1176/appi.ps.201200314. PMID 23584716
- [Background] Weber NS, Cowan DN, Millikan AM, Niebuhr DW. Psychiatric and general medical conditions comorbid with schizophrenia in the National Hospital Discharge Survey. Psychiatr Serv. 2009 Aug;60(8):1059-67. doi: 10.1176/ps.2009.60.8.1059. PMID 19648193
- See also: World Health Organization, 2005. Information Sheet: Premature Death Among People with Mental Illness. — http://www.who.int

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 213 participants were assigned to an arm/group.
Groups:
- Behavioral Weight Loss Intervention: Participants will enroll in the BWLI program for 12 months. BWLI consists of a 8-month initial intervention phase followed by 4-month maintenance phase. The initial intervention phase comprises four types of contact:
  * 1-hour to 1-hour, 30 minute group weight-management class led by facilitator (once per week; 26 classes followed by a one week break and an additional 8 weight management review classes)
  * 45 minute, physical activity led by facilitator (one-two times per week);
  * 20 minute, monthly individual visit with facilitator to address barriers to goals and appropriate skills; and
  * weigh-in during weight management group and individual visits (once each week).
  BWLI: BWLI includes group weight management classes, physical activity classes, individual sessions with a facilitator to address goals and barriers to weight loss, and weigh-ins.
- BWLI & Peer Navigator: Participants randomly assigned to this condition will begin simultaneously with BWLI and run concurrently across the eight months of the intervention. Peer navigators will meet individually and face-to-face with research participants in time and places convenient to the person as needed. Specific practices are determined by the research participant with the peer navigator and may include:
  * partnering with participant on BWLI homework;
  * meeting with participant and BWLI facilitator individually;
  * attending all other health care appointments; and
  * partnering on tasks that arise out of those appointments.
  BWLI & Peer Navigator: Participants receive the BWLI condition and partner with a peer navigator. Peer navigators will meet individually and face-to-face with participants to address their health and weight goals (i.e. working on BWLI homework, attending health care appointments, and facilitating diet and exercise activities).
Period: Cohort 1
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Started (The sum of number of participants who started in Cohorts 1, 2, and 3 = 234 participants initially enrolled) | 41 | 35 | 30
Completed (The sum of number of participants who completed Cohorts 1, 2, and 3 = 213 participants assigned to a group) | 30 | 30 | 30
Not Completed | 11 | 5 | 0
Not completed — Withdrawal by Subject | 11 | 5 | 0
Period: Cohort 2
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Started | 24 | 28 | 27
Completed | 23 | 27 | 27
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Period: Cohort 3
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Started | 17 | 19 | 13
Completed | 16 | 17 | 13
Not Completed | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual) | Total
Number analyzed (Participants) | 69 | 74 | 70 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 66 | 69 | 68 | 203
  >=65 years | 3 | 5 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.93 (10.48) | 52.91 (8.81) | 51.37 (8.55) | 51.4 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 40 | 124
  Male | 25 | 34 | 30 | 89
Race/Ethnicity, Customized [Number; unit: participants] — Identifying as African American was inclusion criteria. Race/Ethnicity listed refers only to participants who identified as any other Race/Ethnicity, in addition to African American. Thus, total percentage is less than 100.
  participants
    American Indian/Alaskan Native | 3 | 3 | 6 | 12
    Asian | 1 | 1 | 0 | 2
    White/Caucasian | 9 | 2 | 4 | 15
    Native Hawaiian/Pacific Islander | 0 | 2 | 1 | 3
    Other | 3 | 2 | 3 | 8
    Hispanic/Latino | 4 | 5 | 1 | 10
    African American | 69 | 74 | 70 | 213
Region of Enrollment [Number; unit: participants]
  United States | 69 | 74 | 70 | 213
SF-36 Subscale: General Health [Mean (Standard Deviation); unit: units on a scale] — From 36-Item Short Form Health Survey. Assess change in participants' health status and health related quality of life. General Health is one of four measure subscales. General Health subscale includes 5 items. Range from 0-100. Higher score indicates better outcome (better health status).
  units on a scale | 60.20 (23.05) | 58.00 (22.11) | 59.13 (22.66) | 58.59 (22.72)
SF-36 Subscale: Bodily Pain [Mean (Standard Deviation); unit: units on a scale] — From 36-Item Short From Health Survey. Assess change in participants' health status and health related quality of life. Bodily Pain is one of four measure subscales. Bodily Pain subscale includes 2 items. Range from 0-100. Higher score indicates better outcomes (better health status, less pain).
  units on a scale | 59.87 (26.25) | 61.94 (28.91) | 59.96 (27.31) | 61.15 (26.90)
SF-36 Subscale: Physical Functioning [Mean (Standard Deviation); unit: units on a scale] — From 36-Item Short From Health Survey. Assess change in participants' health status and health related quality of life. Physical Functioning is one of four measure subscales. Physical Functioning subscale includes 10 items. Range from 0-100. Higher score indicates better outcome (better health status, less physically limited).
  units on a scale | 63.86 (25.07) | 67.00 (26.51) | 69.23 (22.20) | 66.02 (25.69)
SF-36 Subscale: Emotional Well-Being [Mean (Standard Deviation); unit: units on a scale] — From 36-Item Short From Health Survey. Assess change in participants' health status and health related quality of life. Emotional Well-Being is one of four measure subscales. Emotional Well-Being subscale includes 5 items. Range from 0-100. Higher score indicates better outcome (better health status, less limited by emotional issues).
  units on a scale | 63.58 (20.57) | 60.43 (21.17) | 63.43 (23.53) | 62.40 (21.53)
CES-D (Depression) [Mean (Standard Deviation); unit: units on a scale] — Center for Epidemiological Studies Depression Scale. 10 items. Assess change in participants' experienced symptoms of depression. Range from 0 to 60. Higher scores indicate worse outcome (greater depressive symptoms).
  units on a scale | 23.79 (11.87) | 23.67 (10.97) | 21.93 (11.25) | 23.15 (11.24)
RAS-R (Recovery) [Mean (Standard Deviation); unit: units on a scale] — Based on Original Recovery Assessment Scale. RAS-Revised is shorter 24 item scale with individual items representing aspects of recovery to which participants respond on a 5-point agreement scale (1=strongly disagree, 5=strongly agree). Range from 24-120. Higher scores indicate better outcome (better recovery).
  units on a scale | 95.73 (13.81) | 95.32 (12.44) | 98.21 (11.96) | 96.24 (12.61)
QLS (Quality of Life) [Mean (Standard Deviation); unit: units on a scale] — Quality of Life Scale. 6-items assessing how participants feel about different aspects of their lives including as a whole, accomplishments, how they handle problems, family, and activities (1=Terrible, 7=Delighted). Range from 0 to 126. Higher scores indicate better outcome (better quality of life).
  units on a scale | 27.61 (8.12) | 27.00 (6.78) | 27.58 (6.91) | 27.20 (7.35)
WEL (Weight Efficacy Lifestyle) [Mean (Standard Deviation); unit: units on a scale] — Weight Efficacy Lifestyle Questionnaire. 20 items. Assesses participant confidence in resisting eating in some typical eating situations. Items rated on scale from 0=Not confident at all to 9=Very confident. Scores range from 0 to 180. Higher scores indicate better outcome (greater eating self-efficacy).
  units on a scale | 102.83 (38.32) | 99.22 (31.48) | 99.26 (32.35) | 99.99 (33.69)
EES (Emotional Eating) [Mean (Standard Deviation); unit: units on a scale] — Emotional Eating Scale. Assess change in participants' experienced negative emotions and their relationships with desire to eat. 25 items, (0=No desire to eat, 5=Overwhelming urge to eat). Comprised of 3 subscales, added together for a total score. Range from 0 to 125. Higher scores indicate worse outcome (stronger desire to eat).
  units on a scale | 42.14 (23.25) | 43.14 (21.15) | 40.90 (21.15) | 43.00 (21.52)
Healthy Lifestyle Behaviors Total [Mean (Standard Deviation); unit: units on a scale] — Healthy Lifestyle Behaviors. Assess diet and physical activity. 12 items related to diet, physical activity, and receiving support. Responses from 1=Not at all, never to 5=Most of the time, nearly every day. 12 items totaled for one overall score. Range from 0 to 60. Higher scores indicate better outcome (greater frequency of healthy behaviors).
  units on a scale | 34.82 (8.03) | 34.51 (6.56) | 35.16 (7.85) | 34.70 (7.30)
Healthy Lifestyle Behaviors: Physical Activity Subscale [Mean (Standard Deviation); unit: units on a scale] — Physical Activity subscale of Healthy Lifestyle Behaviors. 5 items (1=Not at all, never; 5=Most of the time, nearly every day). Range from 5 to 25.
  Higher score indicates better outcome (greater physical activity).
  units on a scale | 14.86 (4.16) | 14.38 (3.78) | 14.38 (4.06) | 14.54 (4.00)
Healthy Lifestyle Behaviors: Diet Subscale [Mean (Standard Deviation); unit: units on a scale] — Diet subscale of Healthy Lifestyle Behaviors. 6 items (1=Not at all, never; 5=Most of the time, nearly every day). Range from 6 to 30. Higher scores indicate better outcome (greater frequency of healthy diet behaviors).
  units on a scale | 18.12 (4.78) | 18.20 (4.56) | 18.54 (4.87) | 18.29 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Change in Weight (pounds/lbs)
Time Frame: 0, 4, 8 and 12 months
Population: Data collection for Weight variable was challenging (COVID, transition to online) and ultimately discontinued after Cohort 1. The results and intent-to-treat analyses for Weight are based on data from subset of participants before Weight data collection ceased.
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 31 | 28 | 31
pounds (lbs)
  Baseline | 226.54 (41.22) | 225.46 (52.94) | 218.19 (40.41)
  4-Month | 225.63 (42.58) | 223.21 (51.27) | 214.85 (40.99)
  8-Month | 227.66 (42.12) | 223.25 (50.63) | 216.03 (39.62)
  12-Month | 228.86 (41.29) | 222.41 (50.13) | 216.65 (39.54)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Test type: Superiority; p = .025, ANOVA; degrees of freedom = (3, 172); Mean Difference (Net) = 0.36

2. Secondary Outcome: Quality of Life Scale (QLS)
Description: Quality of Life Scale. Assesses life domains including general life, daily activities, and social contact. 6-items assessing how participants feel about different aspects of their lives including as a whole, accomplishments, how they handle problems, family, and activities (1=Terrible, 7=Delighted). Range from 0 to 126. Higher scores indicate better outcome (better quality of life).
Time Frame: 0, 8 months
Population: Analysis was performed on "intention-to-treat." Participants were categorized based on research condition assigned at baseline regardless of BHL or PHN attendance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 69 | 74 | 70
score on a scale
  Baseline | 27.61 (8.12) | 27.00 (6.78) | 27.58 (6.91)
  8-Month | 28.63 (7.69) | 28.53 (6.83) | 29.49 (6.84)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intent-to-treat analyses; Test type: Superiority; p = 0.784, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 0.243
Statistical Analysis 2: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses; Test type: Superiority; p = 0.810, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 0.058

3. Secondary Outcome: Recovery Assessment Scale-Revised (RAS-R)
Description: Based on Original Recovery Assessment Scale. RAS-Revised is shorter 24 item scale with individual items representing aspects of recovery to which participants respond on a 5-point agreement scale (1=strongly disagree, 5=strongly agree).There are five factors (1) personal confidence and hope; (2) willingness to ask for help; (3) goal and success orientation; (4) reliance on others; (5) not dominated by symptoms. Range from 24-120. Higher scores indicate better outcome (better recovery).
Time Frame: 0, 8 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 69 | 74 | 70
score on a scale
  Baseline | 95.73 (13.81) | 95.32 (12.44) | 98.21 (11.96)
  8-Month | 98.72 (14.33) | 98.85 (13.01) | 97.65 (13.92)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intent-to-treat analyses; Test type: Superiority; p = 0.174, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 1.77
Statistical Analysis 2: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses; Test type: Superiority; p = 0.286, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 1.15

4. Secondary Outcome: Weight Efficacy Lifetime (WEL) Questionnaire
Description: Weight Efficacy Lifestyle Questionnaire. 20 items. Assesses participant confidence in resisting eating in some typical eating situations. Items rated on scale from 0=Not confident at all to 9=Very confident. Scores range from 0 to 180. Higher scores indicate better outcome (greater eating self-efficacy).
Time Frame: 0, 8 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 69 | 74 | 70
score on a scale
  Baseline | 102.83 (38.32) | 99.22 (31.48) | 99.26 (32.35)
  8-Month | 124.72 (33.81) | 116.13 (32.40) | 109.93 (39.06)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intent-to-treat analyses; Test type: Superiority; p = 0.261, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 1.36
Statistical Analysis 2: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses; Test type: Superiority; p = 0.912, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 0.012

5. Secondary Outcome: Self-Efficacy for Exercise Scale
Description: Assesses participant beliefs in their ability to continue exercising on a three-time per week basis at moderate intensities. Range from 0 to 90. Higher score = better.
Time Frame: 0, 8 months
Population: Due to COVID-19, interviews were transitioned online to be conducted virtually. In order to minimize participant fatigue, secondary outcome measures including this Self-Efficacy for Exercise Scale were discontinued. The 8 Month values refer to subset of participants who completed 8 Month interview before the Self-Efficacy for Exercise Scale was discontinued.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 62 | 64 | 64
score on a scale
  0 Month | 74.05 (24.50) | 69.02 (23.88) | 76.56 (22.70)
  8 Month: number analyzed (Participants) | 44 | 44 | 39
  8 Month | 66.34 (24.28) | 62.10 (25.62) | 67.15 (23.82)

6. Secondary Outcome: Waist Circumference
Description: Change in waist circumference
Time Frame: 0, 4, 8, 12 months
Population: Data collection for Waist Circumference variable was challenging (COVID, transition to online) and ultimately discontinued after Cohort 1. The results and intent-to-treat analyses for Waist Circumference are based on data from subset of participants before Waist Circumference data collection ceased.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 31 | 28 | 31
inches
  0 Months (Baseline) | 46.00 (4.54) | 43.85 (6.18) | 44.99 (5.61)
  4 Months | 45.56 (4.90) | 44.78 (6.90) | 44.60 (6.34)
  8 Months | 46.23 (4.69) | 44.36 (6.44) | 43.82 (6.16)
  12 Months | 45.98 (5.04) | 44.13 (6.58) | 43.99 (5.59)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Test type: Superiority; p = 0.11, ANOVA; degrees of freedom = 3, 172; Mean Difference (Net) = 1.74

7. Secondary Outcome: Blood Pressure
Description: Mean diastolic and systolic blood pressure (BP), in millimeters of mercury (mmHg) across 4 time frames.
Time Frame: 0, 4, 8, 12 months
Population: Data collection for Blood Pressure variable was challenging (COVID, transition to online) and ultimately discontinued after Cohort 1. The results and intent-to-treat analyses for Blood Pressure are based on data from subset of participants before Blood Pressure data collection ceased.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 27 | 25 | 30
millimeters of mercury (mmHg)
  0 Month (Baseline) Mean systolic BP | 127.39 (15.52) | 124.98 (25.97) | 126.85 (25.79)
  0 Month (Baseline) Mean diastolic BP | 89.11 (13.12) | 92.10 (12.55) | 90.27 (14.23)
  4 Month Mean systolic BP | 129.35 (18.34) | 129.12 (25.78) | 125.93 (15.99)
  4 Month Mean diastolic BP | 87.22 (14.13) | 86.62 (14.54) | 84.50 (10.06)
  8 Month Mean systolic BP | 132.83 (21.30) | 124.80 (21.18) | 125.43 (18.22)
  8 Month Mean diastolic BP | 86.87 (13.79) | 83.20 (12.31) | 85.63 (13.16)
  12 Month Mean systolic BP | 130.06 (19.89) | 133.68 (24.34) | 130.95 (14.02)
  12 Month Mean diastolic BP | 86.70 (13.25) | 87.46 (12.06) | 86.52 (9.26)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Mean systolic blood pressure; Test type: Superiority; p = 0.09, ANOVA; degrees of freedom = 3, 156; Mean Difference (Net) = 1.18
Statistical Analysis 2: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Mean diastolic blood pressure; Test type: Superiority; p = 0.05, ANOVA; degrees of freedom = 3, 156; Mean Difference (Net) = 0.63

8. Secondary Outcome: Height
Description: Measure participants' height (inches)
Time Frame: 0 Month (Baseline)
Population: Physical measurement only collected once (at Baseline)
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 69 | 70 | 74
inches | 65.38 (3.65) | 66.68 (3.85) | 66.29 (4.70)

9. Secondary Outcome: 36-Item Short Form Health Survey (SF-36)
Description: 36-Item Short Form Health Survey. Assess change in participants' health status and health related quality of life. Includes 4 subscales: (1) General health, (2) bodily pain, (3) physical functioning, (4) emotional well-being; range from 0-100 for each subscale. Higher score indicates better outcome.
Time Frame: 0, 8 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 69 | 74 | 70
score on a scale
  0 Month-General Health Subscale (Baseline) | 60.20 (23.05) | 58.00 (22.11) | 59.13 (22.66)
  0 Month-Bodily Pain Subscale (Baseline) | 59.87 (26.25) | 61.94 (28.91) | 59.96 (27.31)
  0 Month-Physical Functioning Subscale (Baseline) | 63.86 (25.07) | 67.00 (26.51) | 69.23 (22.20)
  0 Month-Emotional Well-Being Subscale (Baseline) | 63.58 (20.57) | 60.43 (21.17) | 63.43 (23.53)
  8 Month-General Health Subscale | 62.11 (20.53) | 64.23 (21.96) | 58.17 (24.92)
  8 Month-Bodily Pain Subscale | 58.11 (27.13) | 63.25 (29.94) | 59.52 (26.29)
  8 Month-Physical Functioning Subscale | 59.74 (27.72) | 68.54 (27.23) | 60.48 (28.12)
  8 Month-Emotional Well-Being Subscale | 64.49 (20.70) | 67.20 (18.27) | 68.32 (18.86)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Test type: Superiority — Intention-to-treat analyses. General Health subscale; p = 0.121, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 2.14
Statistical Analysis 2: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses. General Health subscale; Test type: Superiority; p = 0.193, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 1.71
Statistical Analysis 3: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intention-to-treat analyses. Bodily Pain subscale; Test type: Superiority; p = 0.835, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 0.181
Statistical Analysis 4: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses, Bodily Pain subscale; Test type: Superiority; p = 0.513, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 0.430
Statistical Analysis 5: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intention-to-treat analyses, Physical Functioning subscale; Test type: Superiority; p = 0.097, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 2.37
Statistical Analysis 6: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses, Physical Functioning subscale; Test type: Superiority; p = 0.184, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 0.040
Statistical Analysis 7: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intention-to-treat analyses. Emotional Well-Being subscale; Test type: Superiority; p = 0.347, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 1.06
Statistical Analysis 8: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses, Emotional Well-Being subscale; Test type: Superiority; p = 0.549, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 0.361

10. Secondary Outcome: Center for Epidemiologic Studies Depression Scale-Depression(CES-D)
Description: Assess change in participants' experienced symptoms associated with depression. 10 items. Range from 0-60. Higher score indicates worse outcome (greater depressive symptoms).
Time Frame: 0, 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 69 | 74 | 70
score on a scale
  Baseline | 23.79 (11.87) | 23.67 (10.97) | 21.93 (11.25)
  8-Month | 21.04 (12.93) | 20.53 (12.09) | 20.07 (11.22)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intention-to-treat analyses; Test type: Superiority; p = .855, ANOVA; Degrees of freedom = 2,182; Mean Difference (Net) = 0.157
Statistical Analysis 2: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses; Test type: Superiority; p = 0.915, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 0.011

11. Secondary Outcome: Evidence-Based Practices Use (EBPU)
Description: Assess change in participants' enrollment in clinical and service interventions. Range from 0-10, higher scores = better outcome.
Time Frame: 0 months
Population: Due to COVID-19, interviews were transitioned online to be conducted virtually. In order to minimize participant fatigue, secondary outcome measures including this Evidence-Based Practices Use (EBPU) were discontinued.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 68 | 73 | 70
score on a scale | 4.07 (2.46) | 4.21 (2.65) | 4.09 (2.48)

12. Secondary Outcome: Emotional Eating Scale (EES)
Description: Assess change in participants' experienced negative emotions and their relationships with desire to eat. 25 items. (0=No desire to eat, 5=Overwhelming urge to eat). Comprised of 3 subscales, added together for a total score. Range from 0 to 125. Higher scores indicate worse outcome (stronger desire to eat).
Time Frame: 0, 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 69 | 74 | 70
score on a scale
  Baseline | 42.14 (23.25) | 43.14 (21.15) | 40.90 (21.15)
  8-Month | 35.60 (20.58) | 33.63 (21.26) | 36.61 (21.38)
Statistical Analysis 1: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); Intent-to-treat analyses; Test type: Superiority; p = 0.508, ANOVA; degrees of freedom = 2, 182; Mean Difference (Net) = 0.680
Statistical Analysis 2: Comparison: Behavioral Weight Loss Intervention vs BWLI & Peer Navigator vs Integrated Care (Treatment as Usual); As-treated analyses; Test type: Superiority; p = 0.198, ANOVA; degrees of freedom = 1, 118; Mean Difference (Net) = 1.67

13. Secondary Outcome: Life Events Checklist for DSM-5
Description: Life Events Checklist (LEC) for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Assess participants experiences of potential traumatic events on a 6-point nominal scale, across 16 types of traumatic events. No formal scoring protocol or interpretation recommended. Reported scores indicate average amount of distress by traumatic event type. Higher values indicate greater distress from exposure to trauma = worse outcomes (Minimum = 0, maximum = 7).
Time Frame: Baseline
Population: Due to COVID-19, interviews were transitioned online to be conducted virtually. In order to minimize participant fatigue, secondary outcome measures, including this Life Events Checklist for DSM-5 was discontinued. Overall number of participants analyzed refers to those who completed the measure before it was discontinued. Number of participants analyzed in each row endorsed history of that trauma type. There was not enough data collected for further analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
Number analyzed (Participants) | 68 | 73 | 70
score on a scale
  Natural Disaster: number analyzed (Participants) | 13 | 14 | 18
  Natural Disaster | 4.08 (2.53) | 3.71 (2.05) | 2.94 (2.21)
  Fire or Explosion: number analyzed (Participants) | 14 | 21 | 22
  Fire or Explosion | 3.86 (2.21) | 3.52 (2.48) | 3.09 (2.37)
  Transportation Accident: number analyzed (Participants) | 25 | 32 | 22
  Transportation Accident | 4.28 (1.90) | 3.84 (2.49) | 3.09 (2.25)
  Serious Accident at Work/Home/Recreational: number analyzed (Participants) | 16 | 18 | 11
  Serious Accident at Work/Home/Recreational | 4.06 (1.53) | 4.67 (2.54) | 5.36 (1.43)
  Exposure to Toxic Substance: number analyzed (Participants) | 6 | 8 | 10
  Exposure to Toxic Substance | 4.00 (2.97) | 4.88 (2.64) | 5.00 (1.89)
  Physical Assault Without a Weapon: number analyzed (Participants) | 27 | 32 | 25
  Physical Assault Without a Weapon | 4.96 (1.97) | 4.66 (2.43) | 4.24 (2.31)
  Assault With a Weapon: number analyzed (Participants) | 22 | 24 | 26
  Assault With a Weapon | 4.82 (1.97) | 5.04 (2.29) | 3.81 (2.35)
  Sexual Assault: number analyzed (Participants) | 22 | 30 | 26
  Sexual Assault | 5.82 (1.68) | 5.60 (2.31) | 4.73 (2.27)
  Other Unwanted or Uncomfortable Sexual Experience: number analyzed (Participants) | 17 | 19 | 12
  Other Unwanted or Uncomfortable Sexual Experience | 5.12 (1.50) | 5.05 (2.46) | 5.08 (2.47)
  Combat: number analyzed (Participants) | 5 | 2 | 10
  Combat | 2.80 (1.30) | 4.00 (4.24) | 3.30 (2.41)
  Captivity: number analyzed (Participants) | 8 | 6 | 8
  Captivity | 5.62 (2.07) | 5.33 (1.51) | 6.00 (1.31)
  Life-threatening Illness or Injury: number analyzed (Participants) | 22 | 19 | 21
  Life-threatening Illness or Injury | 5.00 (1.80) | 4.63 (2.36) | 4.38 (2.33)
  Severe Human Suffering: number analyzed (Participants) | 17 | 14 | 14
  Severe Human Suffering | 5.41 (1.42) | 5.14 (2.32) | 5.57 (1.79)
  Serious Injury, Harm, or Death Caused: number analyzed (Participants) | 6 | 9 | 9
  Serious Injury, Harm, or Death Caused | 5.67 (1.21) | 3.56 (2.83) | 6.11 (1.36)
  Incarceration: number analyzed (Participants) | 23 | 28 | 27
  Incarceration | 4.52 (2.15) | 3.86 (2.70) | 4.15 (2.49)
  Homelessness: number analyzed (Participants) | 30 | 36 | 32
  Homelessness | 4.60 (2.16) | 5.06 (2.59) | 4.75 (2.34)
  Involuntary Hospitalization: number analyzed (Participants) | 19 | 16 | 17
  Involuntary Hospitalization | 4.26 (2.33) | 3.94 (2.72) | 4.65 (2.18)
  Exposure to Neighborhood Violence: number analyzed (Participants) | 23 | 29 | 30
  Exposure to Neighborhood Violence | 4.61 (2.31) | 4.45 (2.34) | 4.97 (2.00)
  Any Other Very Stressful Event: number analyzed (Participants) | 6 | 11 | 7
  Any Other Very Stressful Event | 6.67 (0.52) | 6.27 (1.27) | 5.71 (1.38)

ADVERSE EVENTS:
Time Frame: 2 years, 11 months
Description: Adverse Event: Any unfavorable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporarily associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research. Severe Adverse Event: Event severity determined by scale, 1 is an adverse event of minimal severity, and 4 is an adverse event of maximal severity:
Arm/Group | Behavioral Weight Loss Intervention | BWLI & Peer Navigator | Integrated Care (Treatment as Usual)
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/74 | 0/70
Serious Adverse Events (participants affected / at risk) | 1/69 | 1/74 | 0/70
Other Adverse Events (participants affected / at risk) | 0/69 | 0/74 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Weight Loss Intervention (N=69) | BWLI & Peer Navigator (N=74) | Integrated Care (Treatment as Usual) (N=70)
High blood pressure observed at interview (General disorders) | 0 (0) | 1 (1) | NA (0) — Participant's blood pressure was observed to be very high during data collection (1st reading: 160+/109) (2nd reading: 150+/109). Research interviewer notified medical team at clinic. Caseworker waited until transfer to hospital for evaluation.
Difficulty walking to interview, back pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Researcher observed participant in hallway. Co-Investigator was consulted & present. 2 public safety officers assisted until participant was picked up by caseworker.

LIMITATIONS AND CAVEATS:
Difficulties with study retention led to missing data, which limited power and options for data analysis. COVID-19 challenges forced a change to online format, impacting standardization of delivery across cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT03382782/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT03382782/ICF_001.pdf